CLINICAL TRIAL: NCT05015985
Title: Benefits of a Music-based Self-relaxing Program Application (MUSIC-CARE) Combined to Locoregional Anesthesia for Forearm Orthopedic Surgery : A Randomized Trial
Brief Title: MUSIC-CARE and Locoregional Anesthesia for Orthopedic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: American Hospital of Paris (Other)
Responsible Party: Principal Investigator, Gilles BOCCARA, principal investigator, American Hospital of Paris
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MUSICARE/ALR/ORTHO1
Record Dates: First submitted 2021-04-24; First posted 2021-08-23 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Regional Anesthesia; Music; Forearm; Injury, Superficial, Multiple (With Elbow)
Keywords: musicotherapy,; anxiety; pain; locoregional anesthesia; orthopedic surgery; Musicare
MeSH Terms: conditions — Wounds and Injuries; Anxiety Disorders; Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: In this study, the investigators compare a specific program of music therapy to an usual music support by playlist. The specific program MUSIC-CARE is administered through a hardware and software, consisting of a modern tablet. The Music-Care app is a receptive music intervention, allowing the patient to freely adjust the length of and choose the preferred style between different sequences of instrumental music. All musical pieces were recorded in high-quality recording studios with professional musicians.
  Music-Care utilizes the "U" technique designed to gradually relax the listener. Initially, the objective is to represent the patient's state of tension by stimulating musical rhythm of 80-95 beats per minute (bpm). Then, it gradually falls into a relaxed state via a gradual reduction in musical tempo (40-80 bpm), orchestral size, frequencies, and volume (descending arm of the "U").
Who Masked: Care Provider, Outcomes Assessor
Masking Description: During all the procedure, the anesthetist performing the locoregional anesthesia and the intravenous hypnotic administration, is blinded about the patient group and music program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MUSIC-CARE Group (Active Comparator): In the Music-Care group, a program of music therapy was administered through a hardware and software provided to the investigative team by the Music-Care Company. The standardized techniques include three sequences in which the relaxing, maintenance and simulating times differ.
  Music-Care utilizes the "U" technique designed to gradually relax the listener. In the current study, music sequences during patients' sessions were based on the mount "U", and instrumental musical works were selected for a varying numbers styles (classical, jazz, world music, etc.) and adapted to the patient's style via patient request.
  Interventions: Other: Music-Care
- CONTROL group (Sham Comparator): In the control group, a music program from an established playlist with various instrumental music is chosen by the patient and delivered by the same tablet.
  Interventions: Other: control group

INTERVENTIONS:
Other: Music-Care — music relaxation by a specific hardware and software program application (MUSIC-CARE)
  Arms: MUSIC-CARE Group
Other: control group — music relaxation using a music playlist supply (control group)
  Arms: CONTROL group

SUMMARY:
Anxiety, fright, stress and pain have always been sources of emotional distress for patients undergoing invasive procedures in clinical settings. Experts have long used traditional methods such as analgesics and anxiolytics to address these issues. But, backed by a movement aiming at reducing the use of pharmacological products, alternative interventions, including music therapy, have gained some steam in recent years. These interventions may have the ability to reduce pain and anxiety while increasing relaxation, coping skills and the overall experience of the procedure. For orthopedic surgery, anesthetics could propose general anesthesia or locoregional anesthesia. The upper limb orthopedic surgery is often performed under locoregional anesthesia and in the ambulatory procedure. However, with the known exacerbating effects of stress and anxiety on pain, the affective experience of the patient can be negatively influenced. In order to mitigate these problems, various types of sedatives and anxiolytics and even low-dose propofol can be used.

The Montpellier Regional University Hospital, along with the Music Care Company developed a software so as to standardize this technique around these recommendations. This model demonstrated its efficacy in both acute and chronic pain settings. Indeed, a single music therapy session was found to be effective for decreasing anxiety and promoting relaxation, as indicated by decreases in heart rate, blood pressure, BIS and respiratory rate over the intervention period in intubated patients during weaning phase. Also, a patient-controlled music intervention administered by Music Care has shown to alleviate negative psychological (e.g., depression) and physiological (e.g., pain and discomfort) outcomes and, very importantly, to reduce the consumption of medication in patients with chronic pain due to lumbar pain, fibromyalgia, inflammatory or neurological diseases.

Given the recent availability of a standardized and proven delivery method of music therapy (i.e. MUSIC-CARE), the principal aim of this randomized clinical trial is to assess the effect of this music therapy program delivered by application compared to usual playlist music on drug consumptions and physiological parameters, pain, anxiety levels in patients undergoing forearm orthopedic surgery under locoregional anesthesia.

DETAILED DESCRIPTION:
This is a randomized controlled clinical study on patients who were followed during their forearm orthopedic surgery. The research has been submitted and approved by the Institutional review Board (IRB) at the American Hospital of Paris. Before their inclusion in the study, after to give their consentment, patients were verbally given details about the methods and techniques of the music session.

Patients scheduled to undergo forearm orthopedic surgery (SR) under regional anesthesia are recruited in this study. They are assigned to one of 2 groups in a randomized manner. Excluding criteria are age less 18 years or up 80 years, patients who do not like music for cultural reason, having serious psychiatric disorder, or with not paired deafness or paired one with devices that were incompatible with wearing a headset. After randomization, patients are placed in the control group, using a music support from playlist, or assigned to the MUSICARE group.

In both group, after per os hydroxyzine premedication, each patient received a regional anesthesia using mepivacaine 2%, at least 20 minutes before skin incision under tourniquet. The regional anesthesia is performed using either an axillary plexus block or mild-arm trunk nerve block with electrical nerve stimulation and ultrasound nerve localization. The music support is started before to do the regional anesthesia and continued during all the orthopedic procedure. According to the anxiety level and patient request, an intravenous titration of midazolam was infused 1 mg per 1 mg to get a sedative score less or equal to 1. If this target is not met after 3 mg of midazolam, the anesthetist could infuse a low dose of propofol (20 mg).

During all the procedure, the anesthetist performing the regional anesthesia and the intravenous hypnotic administration, is blinded about the patient group and musicThe Music-Care app is a receptive music intervention, allowing the patient to freely adjust the length of and choose the preferred style between different sequences of instrumental music. All musical pieces were recorded in high-quality recording studios with professional musicians.

Music-Care utilizes the "U" technique, designed to gradually relax the listener. In the current study, music sequences during patients' sessions were based on the mount "U", and instrumental musical works were selected for a varying numbers styles (classical, jazz, world music, etc.) and adapted to the patient's style via patient request. The "U" technique is implemented using a musical sequence of 20 minutes that was divided into 5 different musical pieces at 3 to 4 minutes each. Initially, the objective is to represent the patient's state of tension by stimulating musical rhythm of 80-95 beats per minute (bpm). From there, the remaining 4 sub-pieces are presented in a blended fashion in an attempt for the patient to gradually fall into a relaxed state via a gradual reduction in musical tempo (40-80 bpm), orchestral size, frequencies, and volume (descending arm of the "U"). The music session then reaches a phase of maximum relaxation (downward phase of the "U") before a phase that gradually returns to baseline dynamics (ascending arm of the "U").

In the control group, a music program from an established playlist with various instrumental music is chosen by the patient and delivered by the same tablet.

program. The primary study end points were the consumptions in sedatives (midazolam and propofol), from 10 minutes prior to the procedure until its end. Secondary study end points were pain and anxiety scores as measured the Numeric Rating Scale (NRS) and the Amsterdam Preoperative Anxiety and Information Scale (APAIS), collected before and right after the end of the procedure in the recovery room. We also evaluated the physiological parameters, such as sedation score ( 0: awake; 1: unconsciousness but reactive to verbal stimulation; 2: unconsciousness but reactive to nociceptive stimulation; 3: areactive to stimulation) , heart rate, arterial blood pressure, oxygen saturation at different time points between T0 (10 minutes prior to the beginning of the procedure) and T45 (45 minutes after it). Satisfaction was also collected using a scale from 0 to 5, with a higher score for a high satisfaction, right after the end of the procedure in the recovery room.

ELIGIBILITY:
Inclusion Criteria:

* scheduled forearm orthopedic surgery
* locoregional anesthesia

Exclusion Criteria:

* age below 18 yrs or up to 80 yrs
* emergency
* surgery duration up to 90 minutes
* patient refusing locoregional anesthesia
* local contreindication to locoregional anesthesia
* patients who do not like music for cultural reason,
* patients having serious psychiatric disorder or cognitive disease
* patients with not paired deafness or paired one with devices that were incompatible with wearing a headset.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-10 (Estimated); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
sedative requirement | during the intraoperative period
  midazolam and/or propofol peroperative consumption in milligramme

SECONDARY OUTCOMES:
anxiety score change | during the intraoperative period
  Numeric Rating scale NRS of anxiety from 0 to 10
pain score change | during the intraoperative period
  Numeric Rating Scale NRS of pain intensity from 0 to 10
sedation score change | during the intraoperative period
  score of sedation from 0 (awake) to 3 (areactive to stimulation)
satisfaction score | in postoperative period
  score of patient satisfaction from 0 to 5

CONTACTS AND LOCATIONS:
Overall Officials: Gilles BOCCARA, MD, PhD, Principal Investigator — American Hospital of Paris
Locations (1):
- American Hospital of Paris, Neuilly-sur-Seine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hole J, Hirsch M, Ball E, Meads C. Music as an aid for postoperative recovery in adults: a systematic review and meta-analysis. Lancet. 2015 Oct 24;386(10004):1659-71. doi: 10.1016/S0140-6736(15)60169-6. Epub 2015 Aug 12. PMID 26277246
- [Background] Guetin S, Ginies P, Siou DK, Picot MC, Pommie C, Guldner E, Gosp AM, Ostyn K, Coudeyre E, Touchon J. The effects of music intervention in the management of chronic pain: a single-blind, randomized, controlled trial. Clin J Pain. 2012 May;28(4):329-37. doi: 10.1097/AJP.0b013e31822be973. PMID 22001666
- [Background] Graff V, Cai L, Badiola I, Elkassabany NM. Music versus midazolam during preoperative nerve block placements: a prospective randomized controlled study. Reg Anesth Pain Med. 2019 Jul 18:rapm-2018-100251. doi: 10.1136/rapm-2018-100251. Online ahead of print. PMID 31320504
- [Background] Fu VX, Oomens P, Sneiders D, van den Berg SAA, Feelders RA, Wijnhoven BPL, Jeekel J. The Effect of Perioperative Music on the Stress Response to Surgery: A Meta-analysis. J Surg Res. 2019 Dec;244:444-455. doi: 10.1016/j.jss.2019.06.052. Epub 2019 Jul 18. PMID 31326711
- [Background] Zengin S, Kabul S, Al B, Sarcan E, Dogan M, Yildirim C. Effects of music therapy on pain and anxiety in patients undergoing port catheter placement procedure. Complement Ther Med. 2013 Dec;21(6):689-96. doi: 10.1016/j.ctim.2013.08.017. Epub 2013 Sep 1. PMID 24280479